CLINICAL TRIAL: NCT01553175
Title: Determination of the Frequency of BRG1 and BRM Loss in Rhabdoid Tumors
Brief Title: Studying Gene Expression in Samples From Patients With Rhabdoid Tumors
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AREN12B5; COG-AREN12B5 (Other: Children's Oncology Group); CDR0000728521 (Other: Clinical Trials.gov); NCI-2012-00705 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-03-10; First posted 2012-03-14 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Brain and Central Nervous System Tumors; Kidney Cancer
Keywords: childhood atypical teratoid/rhabdoid tumor; rhabdoid tumor of the kidney
MeSH Terms: conditions — Central Nervous System Neoplasms; Kidney Neoplasms; Rhabdoid Tumor | interventions — Gene Expression Profiling; Immunohistochemistry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: DNA analysis
Genetic: gene expression analysis
Genetic: mutation analysis
Genetic: protein expression analysis
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and find biomarkers related to cancer. It may also help doctors find better ways to treat cancer.

PURPOSE: This research trial studies gene expression in samples from patients with rhabdoid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine if BRM is silenced in the majority, if not all, rhabdoid tumors by immunohistochemistry in primary tumors.
* To determine if BRG1 is silenced in the majority, if not all, rhabdoid tumors by immunohistochemistry in primary tumors.
* To determine if GATA1 and/or HDAC2 is overexpressed in the same tumors that lack BRM expression.
* To determine if BRM promoter polymorphisms correlate with loss of BRM expression in primary rhabdoid tumors.
* To determine how BRG1 is silenced in primary rhabdoid tumors by sequencing BRG1 exons in genomic DNA derived from frozen samples.

OUTLINE: Archived tumor tissue samples are analyzed for BRM, BRG1, GATA1, and/or HDAC2 expression by immunohistochemistry. BRM- and BRG1-negative samples are also analyzed.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Tumor samples from patients diagnosed with rhabdoid tumors
* Matched frozen tumor tissue from BRG1-negative tumors (preferred) or matched genomic DNA from tumors, 100 ng per tumor from BRG1-negative tumors
* Any source of DNA from BRG1-negative tumors (tumors, blood, etc.)
* Matched frozen tumor tissue from BRM-negative tumors to confirm that BRM is not mutated or altered but rather epigenetically suppressed when lost in rhabdoid tumors

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with rhabdoid tumors
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2012-03; Primary Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Absence or presence BRG1 and BRM expression in rhabdoid tumors
Mechanism of suppression of BRG1 and BRM genes

CONTACTS AND LOCATIONS:
Overall Officials: David Reisman, MD, PhD, Principal Investigator — University of Florida